CLINICAL TRIAL: NCT03737305
Title: Randomised Controlled Clinical Trial of a Temporomandibular Joint Distraction Device for Patients With Articular Disorders Diagnosis
Brief Title: RCT of a Temporomandibular Joint Distraction Device for Patients With Articular Disorders Diagnosis
Acronym: TMJ_Dist
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fonseca, Julio (Individual)
Responsible Party: Principal Investigator, Júlio Fonseca, Doctor (Dentistry); Principal Investigator, Fonseca, Julio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMJ_Distractor
Record Dates: First submitted 2018-11-03; First posted 2018-11-09 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: TMJ Disc Disorder; TMJ Pain; TMJ Sounds on Opening/Closing the Jaw; TMJ - Injury of Meniscus of Temporomandibular Joint
Keywords: TMJ; Disc Displacement; Temporomandibular Disorders; TMJ Distraction Device; TMJ Pain
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial, in a unique investigation center, non-blinded, parallel-group, comparative and interpretive study of the results of clinical use of a TMJ distraction device in patients with diagnosis of Articular Disorders, compared to the traditional method of treatment using manual physiotherapy.
Who Masked: Outcomes Assessor
Masking Description: The Outcomes Assessor, or secondary investigator does nor have the knowlegde of the group of patients that is being evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Control group of conventional therapy with manual distraction performed by the physiotherapist in the office (active comparator)
  Interventions: Device: Conventional Physical Therapy
- Distractor Test Group (Experimental): Test group with manual distraction performed by the physiotherapist in the office and the condylar distraction performed by the patient with the condylar distraction device in an ambulatory basis.
  Interventions: Device: TMJ Condilar Distraction Device

INTERVENTIONS:
Device: TMJ Condilar Distraction Device — The patients will perform condylar distraction with the condylar distraction device in an ambulatory basis.
  Arms: Distractor Test Group
Device: Conventional Physical Therapy — Conventional Physical Therapy, performed in office by a experienced physical therapist for the TMJ condition.
  Arms: Control Group

SUMMARY:
Articular Disc Displacements are the most common TMJ arthropathy and the articular distraction technique is one of the most common therapeutic resources. It is a technique almost exclusively performed by the physiotherapist and / or dentist, with repeated applications over an extended period of treatment, that can reach several weeks or months, difficult to perform manually by the patient on an ambulatory basis. Currently there are no ambulatory mandibular exercise devices that aim to execute articular distraction. Thus, the objective of this work was to study, design and develop a device capable of performing and / or assisting patients in the articular distraction maneuver.

DETAILED DESCRIPTION:
Temporomandibular disorders are considered a heterogeneous group of psychophysiological disorders of the stomatognathic system (Okeson 1985, Okeson 1993) covering a broad spectrum of muscular, skeletal or both, clinical problems (Nagamatsu-Sakaguchi, Minakuchi et al). They are often initiated by pain, joint sounds and limited function / mandibular movement, and are considered one of the main causal factors of non-dental orofacial pain (Rossetti et al., 2008, Makino, Masaki et al.; Magnusson 1999). Conservative and non-invasive treatment is considered as the one of choice at an early stage, since the symptomatology is usually reduced through the combined use of occlusal appliences, physiotherapy and medication. (De Leeuw, American Academy of Orofacial Pain et al., 2008) The dislocations of the articular disc are the most common arthropathy and are characterized by several stages of clinical dysfunction involving an abnormal interrelationship of the disc condyle complex (more often an anterior or anteromedial disc displacement) (Isberg-Holm and Westesson 1982 ). Pain (in acute cases), changes in mandibular movement pattern and joint noise are the most frequent symptoms.

The causes of disc displacements are not completely established. It has been postulated that, in most cases, the elongation or rupture of the condyle-disc ligaments allows displacement of the disc. (Stegenga, de Bont et al., 1991) Changes in lubrication and synovial fluid quality have also been suggested as possible etiological agents (Nitzan 2001). The presence of osteoarthritis may also precipitate changes in the condyle-disc complex. (De Leeuw, American Academy of Orofacial Pain et al., 2008) In addition to the intervention of the dentist with occlusal appliance (among other resources), mandibular physiotherapy aims to reduce musculoskeletal pain, promote muscle relaxation, reduce muscle hyperactivity, improve muscle control and function, and maximize joint mobility . In addition to the electrotherapeutic means there are several manual therapy techniques directed to TMJ that aim the joint decompression, fibrosis reduction and adhesions at the level of structures such as ligaments or joint capsule, recaptation of the articular disc or adaptation of the retrodiscal tissues. We are talking about intraoral techniques such as condylar distraction or specific exercises of joint mobility or muscle strengthening. (Craane, Dijkstra et al., 2012) In the specific case of joint disc displacements, the condylar distraction technique is one of the most used therapeutic resources. It is a technique that aims to increase the space between the mandibular condyle and the joint fossa of the temporal, decompressing the joint and promoting the adaptation of the articular tissues and / or the disc reuptake. It is a technique almost exclusively performed by the physiotherapist and / or dentist, with repeated applications over an extended period of treatment that can reach several weeks or months, difficult to perform by the patient at home (De Leeuw, American Academy of Orofacial Pain et al, 2008). There are currently only ambulatory mandibular exercise devices that aim to increase the range of mandibular movement through rotation, rototranslation, and condylar translation (eg, TheraPace Jaw Motion Rehab System, TheraPacer Jaw CPM ). None of these devices distracts the joint, so in cases of acute displacement of the disc, with the presence of retrodiscal pain, they may even be counterproductive. Thus, the development of an apparatus capable of performing or assisting patients in the condylar distraction maneuver could prove to be a valuable aid in the treatment of these conditions, increasing patient adherence and reducing costs related to a long treatment time.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a minimum of 18 years of age
2. Diagnosis by the Research Diagnostic criteria of Temporomandibular Disorders (RDC / TMD), of disk displacement with or without reduction, with or without opening limitation (Group IIa, IIb or IIc) and atralgia (Group IIIa)
3. Clinical indication for the proposed treatment

Exclusion Criteria:

1. Patients <18 years
2. Pregnant patients
3. Absence of posterior teeth (not rehabilitated), advanced periodontal disease in the posterior teeth or patients with total dentures that compromise the use of the device
4. Diagnosis by the Research Diagnostic criteria of Temporomandibular Disorders (RDC / TMD), of Osteoarthritis (Group IIIb) and Osteoarthrosis (IIIc)
5. Presence of contralateral TMJ pathology, with no clinical indication for the proposed treatment, limiting the patient's mandibular mobility and influencing patient rehabilitation (eg, ankylosis or myofibrotic contracture)
6. History of surgery at the ATM
7. Patients with systemic disease that may affect the TMJ
8. Aphasia, dementia, or known psychiatric or physical comorbidity that may interfere with communication or compliance during the rehabilitation process.
9. Patients blind, illiterate or with reduced cognitive abilities that may interfere with communication or compliance during the rehabilitation process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of Pain at Rest (Visual Analogic Scale from 0-10) | 0 day, 7 days, 14 days, 28 days and 90 days of the study
  Mandibular Pain at Rest evaluated in a 0-10 (VAS) Visual Analogic Scale being 0 ´´No pain´´ and 10 ´´The worst pain ever´´
Change of Pain in Function (Visual Analogic Scale from 0-10) | 0 day, 7 days, 14 days, 28 days and 90 days of the study
  Mandibular Pain in Function evaluated in a 0-10 (VAS) Visual Analogic Scale being 0 ´´No pain´´ and 10 ´´The worst pain ever´´
Change of Subjective chewing efficiency | 0 day, 7 days, 14 days, 28 days and 90 days of the study
  Subjective chewing efficiency (evaluated in a 0-10 Visual Analogic Scale with 0 being ´´the worst efficiency ever´´ and 10 ´´the best efficiency ever´´)

SECONDARY OUTCOMES:
Change in the Perceived subjective treatment effectiveness | 0 day, 7 days, 14 days, 28 days and 90 days of the study
  Perceived subjective treatment effectiveness on a five-point scale with 0 being ´´no perceived effectiveness´´ and 4 being the ´´maximum effectiveness´´
Change of Jaw range of motion function in millimetres | 0 day, 7 days, 14 days, 28 days and 90 days of the study
  Jaw range of motion function in millimetres (with no pain, with pain and maximum oppening)

CONTACTS AND LOCATIONS:
Overall Officials: Júlio Fonseca, Principal Investigator — Dr.
Locations (1):
- OrisClinic - Júlio Fonseca, Coimbra, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
All the results and further perspectives.